CLINICAL TRIAL: NCT03332316
Title: Effect of Perineural Dexamethasone on the Duration of Popliteal Nerve Block for Anesthesia After Ankle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R17104M; 2017-002185-51 (EudraCT Number)
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain; Nerve Block
MeSH Terms: conditions — Pain, Postoperative | interventions — dexamethasone 21-phosphate; Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DEXA0 (Placebo Comparator): Ropivacaine Hydrochloride Inj 2mg/ml 20 ml and Sodium Chloride 9mg/mL 1 ml perineurally
  Interventions: Drug: Ropivacaine Hydrochloride Inj 2 mg/ml; Drug: Sodium Chloride 9mg/mL
- DEXA1 (Experimental): Ropivacaine Hydrochloride Inj 2 mg/ml 20 ml and Dexamethasone Sodium Phosphate 5mg/ml 0,2 ml and Sodium Chloride 9mg/mL 0,8 ml perineurally
  Interventions: Drug: Dexamethasone Sodium Phosphate; Drug: Ropivacaine Hydrochloride Inj 2 mg/ml; Drug: Sodium Chloride 9mg/mL
- DEXA2 (Experimental): Ropivacaine Hydrochloride Inj 2 mg/ml 20 ml and Dexamethasone Sodium Phosphate 5mg/ml 0,4 ml and Sodium Chloride 9mg/mL 0,6 ml perineurally
  Interventions: Drug: Dexamethasone Sodium Phosphate; Drug: Ropivacaine Hydrochloride Inj 2 mg/ml; Drug: Sodium Chloride 9mg/mL
- DEXA4 (Experimental): Ropivacaine Hydrochloride Inj 2 mg/ml 20 ml and Dexamethasone Sodium Phosphate 5mg/ml 0,8 ml and Sodium Chloride 9mg/mL 0,2 ml perineurally
  Interventions: Drug: Dexamethasone Sodium Phosphate; Drug: Ropivacaine Hydrochloride Inj 2 mg/ml; Drug: Sodium Chloride 9mg/mL

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate — Dexamethasone injection
  Other Names: Oradexon
  Arms: DEXA1; DEXA2; DEXA4
Drug: Ropivacaine Hydrochloride Inj 2 mg/ml — Ropivacaine injection
Drug: Sodium Chloride 9mg/mL — Sodium Chloride injection
  Other Names: Saline

SUMMARY:
Effect of perineural dexamethasone on the duration of popliteal nerve block after ankle/foot surgery

DETAILED DESCRIPTION:
This study is proposed to explore the effect of perineural dexamethasone on the duration of popliteal nerve block for analgesia after ankle surgery.

After ankle or foot arthrodesis patients need a good analgesia. Nevertheless early mobilisation and discharge are important for the healing process after surgery. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe. Perineural dexamethasone added to local anesthetic prolongs the duration of analgesia of the perineural nerve block.

The perineural use of dexamethasone is still off-label. There is a ongoing discussion of which has better benefits, intravenous or perineural dexamethasone.

There are multiple research where the intravenous and perineural dexamethasone use has compared, but there is still a limited amount of research of low dose perineural dexamethasone versus intravenous dexamethasone.

In this study investigators compare different doses of perineural dexamethasone added to ropivacaine 2 mg/ml 20ml. After arthrodesis under spinal anaesthesia the patients receive popliteal block ropivacaine 2 mg/ml 20 ml and dexamethasone of different doses. Groups 1 to 4 has dexamethasone doses 0, 2mg, 3mg or 4 mg.

After the popliteal nerve block investigators follow postoperative pain, opiate consumption, mobilisation and long term quality of life.

Investigators goal is to find a dexamethasone dose which is as low as possible but at the same time covers the need for a good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Adult people under ankle/foot arthrodesis as a curative therapy of ankle arthrosis or situation after ankle injury or malposition

Exclusion Criteria:

Age under 18 years Complicated diabetes mellitus Lack of finnish language skill and/or co-operation Chronic pain Steroid medication in regular use

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
First need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opiate consumption | 48 hours
  Total opiate consumption after surgery
Pain | postoperatively: at 4 hours, at 8 hours,at 12 hours, at 16 hours, at 20 hours, at 24 hours, at 28 hours, 32 hours, at 36 hours, at 40 hours, at 44 hours, at 48 hours,seventh postoperative day
  Numeric rating scale NRS 0-10
Mobilisation | postoperatively: at 4 hours, at 8 hours,at 12 hours, at 16 hours, at 20 hours, at 24 hours, at 28 hours, 32 hours, at 36 hours, at 40 hours, at 44 hours, at 48 hours
  Toe movement every 4 hour during hospitalization
Blood glucose | postoperatively: at 4 hours, at 8 hours,at 12 hours, at 16 hours, at 20 hours, at 24 hours
  Blood glucose every 4 hour during hospitalization

OTHER OUTCOMES:
Quality of life (EQ-5D-3L) -query | Before operation and 6-8 weeks, 6 months, 12 months postoperatively
McGill -pain query | Before operation and 6-8 weeks, 6 months, 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Maija-Liisa Kalliomäki, PhD, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No